CLINICAL TRIAL: NCT03439254
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Obeticholic Acid in Subjects With Compensated Cirrhosis Due to Nonalcoholic Steatohepatitis
Brief Title: Study Evaluating the Efficacy and Safety of Obeticholic Acid in Subjects With Compensated Cirrhosis Due to Nonalcoholic Steatohepatitis
Acronym: REVERSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 747-304
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Compensated Cirrhosis; Nonalcoholic Steatohepatitis
Keywords: Compensated Cirrhosis; Nonalcoholic Steatohepatitis; Fatty Liver Disease; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Obeticholic Acid (OCA) 10 mg (Experimental): 10 mg OCA for up to 18 months
  Interventions: Drug: Obeticholic acid (10 mg)
- Obeticholic Acid (OCA) 10 mg to 25 mg (Experimental): 10 mg OCA for the first 3 months and then may titrate up to 25 mg OCA for the remaining 15 months of the study
  Interventions: Drug: Obeticholic acid (10 mg to 25 mg)
- Placebo (Placebo Comparator): Placebo for up to 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic acid (10 mg) — Tablets administered orally once daily.
  Other Names: OCA; 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
  Arms: Obeticholic Acid (OCA) 10 mg
Drug: Obeticholic acid (10 mg to 25 mg) — Tablets administered orally once daily.
  Other Names: OCA; 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
  Arms: Obeticholic Acid (OCA) 10 mg to 25 mg
Drug: Placebo — Tablets administered orally once daily.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate whether obeticholic acid (OCA; INT-747) can lead to histological improvement in fibrosis with no worsening of NASH in adults with compensated cirrhosis due to NASH.

ELIGIBILITY:
Key inclusion criteria:

1. Subjects with a confirmed diagnosis of NASH and a fibrosis score of 4 based upon the NASH CRN scoring system determined by central reading

Key exclusion criteria:

1. Current or past history of a clinically evident hepatic decompensation event, such as ascites, hepatic encephalopathy (HE), or variceal bleeding
2. Current or past history of CP score ≥7 points
3. Model for End-stage Liver Disease (MELD) score > 12
4. ALT ≥ 5 X ULN
5. Calculated creatinine clearance <60mL/min using Cockcroft-Gault method
6. Hemoglobin A1c (HbA1c) ≥ 9.5 %
7. Evidence of other known forms of chronic liver disease such as alcoholic liver disease, hepatitis B, hepatitis C, PBC, PSC, autoimmune hepatitis, Wilson disease, iron overload, alpha-1-antitrypsin deficiency, drug-induced liver injury, known or suspected hepatocellular carcinoma (HCC)
8. History of liver transplant, or current placement on a liver transplant list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (192):
- United States (120):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Objective GI d/b/a North Alabama GI Research Center, Madison, Alabama
  - Arizona Liver Health, Chandler, Arizona
  - Arizona Liver Health, Glendale, Arizona
  - The Institute for Liver Health, Tucson, Arizona
  - Liver Wellness Center, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - University of California, San Francisco-Fresno, Fresno, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - eStudySite, La Mesa, California
  - Keck Hospital of USC, Los Angeles, California
  - Cedars-Sinani Medical Center, Los Angeles, California
  - Palmtree Clinical Research, INC., Palm Springs, California
  - Stanford University Medical Center, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - Hi Tech and Global Research LLC, Coral Gables, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - UF Health Jacksonville-Gastroenterology Emerson, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Guardian Angel Research Center, INC, Tampa, Florida
  - Florida Medical Clinic, P.A, Zephyrhills, Florida
  - Summit Clinical Research, LLC, Athens, Georgia
  - The Emory Clinic (TEC), Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Aquiant Research, New Albany, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - University of Louisville, Clinical Trials Unit, Louisville, Kentucky
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - UMass Memorial Health Care, Worcester, Massachusetts
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinical Research Center, Wyoming, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Southern Therapy and Advanced Research (STAR) LLC, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CHI Health Alegent Creighton Clinic, Omaha, Nebraska
  - Sierra Clinical Research, Las Vegas, Nevada
  - Amici GI-LLC, Martinsville, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - University at Buffalo, Clinical and Translational Research Center, Buffalo, New York
  - Ichan School of Medicine at Mount Sinai Beth Israel, New York, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - University of North Carolina at Chapel Hill, School of Medicine, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolinas Center for Liver Disease/Carolinas HealthCare System, Huntersville, North Carolina
  - Carolinas Health Care System Center for Liver Disease, Huntersville, North Carolina
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Dayton Gastroenterology, Inc., Beavercreek, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - The Pennsylvania State University and the Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - UPMC - Center for Liver Diseases at the Thomas E. Starzl Institute, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Ralph H. Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - SCTR Research Nexus, Charleston, South Carolina
  - Rapid City Medical Center LLP, Rapid City, South Dakota
  - Gastro One, Germantown, Tennessee
  - Associates in Gastroenterology, PLC, Hermitage, Tennessee
  - Johnson City Medical Center, Johnson City, Tennessee
  - Methodist Healthcare University Hospital, Memphis, Tennessee
  - Quaility Medical Research, PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center - Digestive Disease Center, Nashville, Tennessee
  - Texas Clinical Research Institute LLC, Arlington, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - Texas Digestive Disease Consultants, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Baylor Scott and White All Saints Medical Center, Fort Worth, Texas
  - Texas Digestive Disease Consultants, Fort Worth, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
  - Centex Studies, Inc., McAllen, Texas
  - American Research Corporation, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Texas Digestive Disease Consultants, San Marcos, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Maryview Hospital, Inc. d/b/a Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Richmond Community Hospital, Inc. d/b/a Bon Secours, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Gastroenterology Consultants of Southwest Virginia, Roanoke, Virginia
  - Virginia Mason - Seattle Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Australia (7):
  - Nepean Blue Mountains Local Health District, Nepean Hospital, Kingswood, New South Wales
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - St Vincent's Hospital, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (9):
  - University of Calgary Liver Unit (Heritage Medical Research Clinic), Calgary, Alberta
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Nova Scotia Health Authority, Halifax, Nova Scotia
  - Kent Place, Lindsay, Ontario
  - London Health Sciences Centre-University Hospital, London, Ontario
  - Office of Dr. Gauthier, North Bay, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Clinique de medecine Urbaine du Quartier Latin, Montreal, Quebec
  - Chronic Viral Illness/McGill University Health Centre (MUHC), Montreal, Quebec
- France (13):
  - CHU Amiens Picardie, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital Beaujon- Service d'Hepatologie, Clichy
  - Center Hospitalier Universitaire Grenoble Alpes, La Tronche
  - Hôpital de la Croix Rousse, Lyon
  - CHU de Nice, Hôpital de l'Archet 2, Nice
  - Hôpital Pitié-Salpêtrierè, Paris
  - CHU de Rouen-Centre Hospitalier Universitaire, Rouen
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - Hôpital Hautepierre, Strasbourg
  - Hôpital Purpan, Toulouse
  - CHRU de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse, Villejuif
- Germany (8):
  - Univeritätsklinkum Würzburg, Würzburg, Bavaria
  - Teuber Consulting & Research UG, Frankfurt am Main, Hesse
  - Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - EUGASTRO GmbH, Leipzig, Saxony
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
  - Gastroenterologisch-Hepatologisches Zentrum Kiel, Kiel, Schleswig-Holstein
  - Charité - Universitätsmedzin Berlin, Berlin
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Hungary (3):
  - Synexus Magyarország Kft. Budapest, Budapest
  - Synexus Magyarorszag Kft. Debrecen A.S., Debrecen
  - Synexus Magyarorszag Kft. Gyula DRS, Gyula
- New Zealand (4):
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Public Hospital, Dunedin
  - Wellington Regional Hospital, Wellington
- Poland (8):
  - Synexus Polska Sp. z o.o., Oddział w Częstochowie, Częstochowa
  - Synexus Polska Sp. z.o.o., Oddział w Gdańsku, Gdansk
  - Synexus Polska Sp. Z.o.o., Oddział w Gdyni, Gdynia
  - Synexus Polska Sp. z o.o., Oddział w Katowicach, Katowice
  - Synexus Polska Sp. z o.o., Oddział w Łodzi, Lodz
  - Synexus Polska Sp. z o.o., Oddział w Poznaniu, Poznan
  - Synexus Polska Sp. z o.o., Oddział w Warszawie, Warsaw
  - Synexus Polska Sp. z o.o., Oddział w Wrocławiu, Wroclaw
- Puerto Rico (2):
  - Latin Clinical Trial Center, San Juan
  - Fundación de Investigación de Diego, San Juan
- Spain (7):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politécnic La Fe, Valencia
- Ukraine (2):
  - Medical Center of LLC Medbud-Clinic, Clinical Diagnostic Department, Kyiv
  - Kyiv Railway Clinical Hospital №2 of branch "Health Center" of the Joint-Stock Company "Ukranian Railway", Day treatment department, Kyiv
- United Kingdom (9):
  - Derby Teaching Hospitals NHS Foundation Trust, Derby, Derbyshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Royal Free Hospital NHS Foundation Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, St Mary's Hospital, London, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Derriford Hospital, Plymouth, England
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Freeman Hospital, Newcastle upon Tyne, Tyne and Wear

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a total of around 286 centers.
Pre-assignment Details: This was a Phase 3, double-Blind, randomized, placebo-controlled, multicenter study to evaluate the efficacy and safety of Obeticholic Acid (OCA) in participants with compensated cirrhosis due to Nonalcoholic Steatohepatitis (NASH). The study comprised of a double-blind (DB) phase (18 months) followed by Open-label extension (OLE) phase (12 months).
Groups:
- DB: Placebo: Participants were randomized to receive placebo once daily orally with water, in conjunction with local standard of care.
- DB: OCA 10 Milligrams (mg): Participants were randomized to receive OCA 10 mg once daily dosing orally with water, in conjunction with local standard of care.
- DB: OCA 10 mg Titrated to OCA 25 mg: Participants were randomized to receive OCA 10 mg for the first 3 months prior to uptitrating to OCA 25 mg at Month 3, once daily dosing orally with water, in conjunction with local standard of care. Uptitration was determined based on the laboratory criteria and safety and tolerability assessments completed prior to Month 3. If uptitration at Month 3 was not feasible, the window for uptitration was extended by up to one calendar month, after consultation and agreement with the Medical Monitor.
- OLE: OCA 10 mg (DB Placebo): Participants who completed the DB phase (and continued to receive investigational product) were eligible to enroll into the OLE phase. All participants received OCA upon entry into the OLE phase. Participants randomized to placebo in the DB phase were re-randomized to either receive OCA 10 mg or titrated dose of OCA 25 mg. Uptitration was determined based on the same criteria and assessments as employed in the DB phase.
- OLE: OCA 10 mg (DB OCA 10 mg): Participants who completed the DB phase (and continued to receive investigational product) were eligible to enroll into the OLE phase. All participants received OCA upon entry into the OLE phase. Participants randomized to OCA 10 mg during the DB phase continued the same dosing regimen they received at the end of the DB Phase; however, they underwent dummy titration to maintain study blind until all participants completed the DB phase.
- OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg): Participants who completed the DB phase (and continued to receive investigational product) were eligible to enroll into the OLE phase. All participants received OCA upon entry into the OLE phase. Participants randomized to OCA 10 mg to 25 mg titration during the DB phase continued the same dosing regimen they received at the end of the DB Phase; however, they underwent dummy titration to maintain study blind until all participants completed the DB phase.
Period: Double-blind Phase (18 Months)
Arm/Group | DB: Placebo | DB: OCA 10 Milligrams (mg) | DB: OCA 10 mg Titrated to OCA 25 mg | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Started | 313 | 296 | 310 | 0 | 0 | 0
Completed | 284 | 274 | 275 | 0 | 0 | 0
Not Completed | 29 | 22 | 35 | 0 | 0 | 0
Not completed — Adverse Event | 11 | 12 | 15 | 0 | 0 | 0
Not completed — Covid-19 Non Adverse Event (AE) Related Issues | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 5 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant moved to Kansas | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Site cover and participant was not willing to be transferred | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Stopped Investigational product (IP) due to an AE in Australia | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Drug Holiday | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Spouse underwent surgery and participant was unable to take IP regularly | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Site closure | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 6 | 9 | 0 | 0 | 0
Period: Open Label Extension Phase (12 Months)
Arm/Group | DB: Placebo | DB: OCA 10 Milligrams (mg) | DB: OCA 10 mg Titrated to OCA 25 mg | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Started | 0 | 0 | 0 | 231 | 221 | 207
Completed | 0 | 0 | 0 | 215 | 208 | 192
Not Completed | 0 | 0 | 0 | 16 | 13 | 15
Not completed — Adverse Event | 0 | 0 | 0 | 8 | 5 | 7
Not completed — Bariatric Surgery | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Covid-19 Non-AE Related Issues | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Increase CR from Baseline | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Medical reasons by Sponsor | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) Population: included all randomized participants.
Groups:
- DB: OCA 10 mg Titrated to OCA 25 mg: Participants were randomized to receive OCA 10 mg for the first 3 months prior to uptitrating to OCA 25 mg at Month 3, once daily dosing orally with water, in conjunction with local standard of care. Uptitration was determined based on the laboratory criteria and safety and tolerability assessments completed prior to Month 3. If uptitration at Month 3 was feasible, the window for uptitration was extended by up to one calendar month, after consultation and agreement with the Medical Monitor.
- Total: Total of all reporting groups
Arm/Group | DB: Placebo | DB: OCA 10 Milligrams (mg) | DB: OCA 10 mg Titrated to OCA 25 mg | Total
Number analyzed (Participants) | 313 | 296 | 310 | 919
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (8.99) | 60.1 (8.70) | 60.1 (8.67) | 59.9 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 184 | 209 | 605
  Male | 101 | 112 | 101 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 52 | 55 | 151
  Not Hispanic or Latino | 246 | 217 | 233 | 696
  Unknown or Not Reported | 23 | 27 | 22 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 4 | 10
  Asian | 8 | 5 | 5 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 3 | 4
  Black or African American | 4 | 6 | 4 | 14
  White | 272 | 254 | 272 | 798
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 25 | 25 | 21 | 71

OUTCOME MEASURES:

1. Primary Outcome: DB Phase: Number of Participants Who Were Responders and Showed Improvement in Fibrosis by at Least 1 Stage Without Worsening of Nonalcoholic Steatohepatitis (NASH)
Description: Fibrosis stage was evaluated by NASH Clinical Research Network(CRN)Fibrosis Staging System with stages:0=no fibrosis;1=perisinusoidal/periportal;1A=mild,zone 3,perisinusoidal;1B=moderate,zone 3,perisinusoidal;1C=portal/periportal;2=perisinusoidal and portal/periportal;3=bridging fibrosis;4=cirrhosis.No worsening of steatohepatitis was defined as no worsening of lobular inflammation or hepatocellular ballooning grade as per scoring in relevant nonalcoholic fatty liver disease activity score (NAS) categories.NAS is semiquantitative scoring system based on unweighted sum of:steatosis (0=<5% to 3=>66%),lobular inflammation(0=no foci to 3=>4 foci/200x),hepatocellular ballooning(0=none to 2=many cells/prominent ballooning)scores.Total scale range:0-12;0:no features of fatty liver disease and 12:highest degree of fatty liver disease.Higher scores:worse symptoms.Responders:did not discontinue treatment due to Adverse event(AE) or did not die and had evaluable post-Baseline biopsy assessment
Time Frame: Up to 18 months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB: Placebo | DB: OCA 10 Milligrams (mg) | DB: OCA 10 mg Titrated to OCA 25 mg
Number analyzed (Participants) | 313 | 296 | 310
Participants | 31 | 33 | 37
Statistical Analysis 1: Comparison: DB: Placebo vs DB: OCA 10 Milligrams (mg); Test type: Other; p = 0.6172, Cochran-Mantel-Haenszel; Response ratio(Mantel-Haenszel estimate) = 1.13, 95% CI 2-sided [0.71 to 1.79] — Treatment / Placebo Response Ratio = Percentage of Responders in Active Treatment Arm / Percentage of Responders in Placebo, stratified by Baseline diabetes status (yes/no)
Statistical Analysis 2: Comparison: DB: Placebo vs DB: OCA 10 mg Titrated to OCA 25 mg; Test type: Other; p = 0.4184, Cochran-Mantel-Haenszel; Response ratio(Mantel-Haenszel estimate) = 1.20, 95% CI 2-sided [0.77 to 1.89] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: OLE Phase: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to 12 months
Population: Safety Population: included all randomized participants who received at least 1 dose of investigational product (OCA or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Number analyzed (Participants) | 231 | 221 | 207
Participants
  AEs | 199 | 213 | 197
  SAEs | 26 | 50 | 48

3. Primary Outcome: OLE Phase: Change From Baseline to Month 12 in Liver Stiffness Measurement (LSM)
Description: Non-invasive radiological methods to assess liver stiffness were conducted at selected study sites where the respective devices were available. These assessments were taken by vibration controlled transient elastography (TE) method using FibroScan®. Participant was included as a random effect and an unstructured covariance matrix was used assuming convergence could be attained. Baseline was defined as the last value collected prior to the first administration of the investigational product (IP). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Month 12
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Kilopascal (kPa)
Arm/Group | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Number analyzed (Participants) | 177 | 172 | 160
Kilopascal (kPa) | -2.10 [-7.40 to 3.40] | -2.90 [-7.75 to 1.35] | -3.45 [-7.85 to 0.75]

4. Primary Outcome: OLE Phase: Fibrosis-4 (FIB-4) at Baseline
Description: FIB-4 was a noninvasive assessment of liver disease assessed by a combination of age, alanine aminotransferase (ALT) and platelet results. FIB-4 was the ratio of age in years and aminotransferase to platelet count. It was a non-invasive hepatic fibrosis index score combining standard biochemical values, platelets, ALT, Aspartate aminotransferase (AST) and age that was calculated using formula: FIB-4 = (Age [years] x AST [Units per Liter {U/L}]) / (platelets [10^9/L] x (square root of ALT [U/L])). A FIB-4 index of <1.45 indicated no or moderate fibrosis and an index of > 3.25 indicated extensive fibrosis/cirrhosis. Higher ratio indicated worse condition. Baseline was defined as the last value collected prior to the first administration of the IP.
Time Frame: Baseline (Day 1)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Number analyzed (Participants) | 230 | 221 | 207
Ratio | 2.179 (1.0342) | 2.267 (0.9567) | 2.266 (1.0867)

5. Primary Outcome: OLE Phase: Enhanced Liver Fibrosis (ELF) at Baseline
Description: ELF was non-invasive panel of circulating fibrosis markers calculated from serum biomarkers. The markers of fibrosis comprised hyaluronic acid (HA), tissue inhibitor of metalloproteinase (TIMP1) and procollagen III N-terminal peptide (PIIINP). Each of these markers was measured by an immunoassay and an ELF score was generated, from which a level of fibrosis severity could be determined. The ELF test was a composite score: < 7.7: no to mild fibrosis; ≥ 7.7 - < 9.8: Moderate fibrosis; ≥ 9.8 - < 11.3: Severe fibrosis; ≥ 11.3: Cirrhosis.; higher ELF scores were associated with worsening liver fibrosis. Baseline was defined as the last value collected prior to the first administration of the IP.
Time Frame: Baseline (Day 1)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Number analyzed (Participants) | 227 | 220 | 206
Scores on a scale | 10.46 (0.933) | 10.50 (0.940) | 10.48 (0.821)

6. Primary Outcome: OLE Phase: Number of Participants Reporting All-cause Mortality
Description: All-cause mortality is defined as death due to any cause. Number of participants reporting all-cause mortality is presented
Time Frame: Up to Month 12
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Number analyzed (Participants) | 231 | 221 | 207
Participants | 1 | 0 | 1

7. Secondary Outcome: DB Phase: Change From Baseline to Month 18 in LSM
Description: Non-invasive radiological methods to assess liver stiffness were conducted at selected study sites where the respective devices were available. These assessments were taken by vibration controlled TE method using FibroScan®. Participant was included as a random effect and an unstructured covariance matrix was used assuming convergence could be attained. The principal comparison was at Month 18. Baseline was defined as the last value collected prior to the first administration of the IP. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Month 18
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Kilopascal (kPa)
Arm/Group | DB: Placebo | DB: OCA 10 Milligrams (mg) | DB: OCA 10 mg Titrated to OCA 25 mg
Number analyzed (Participants) | 189 | 174 | 173
Kilopascal (kPa) | -0.50 [-5.20 to 5.60] | -3.10 [-7.30 to 3.20] | -2.90 [-8.10 to 2.50]

8. Secondary Outcome: DB Phase: FIB-4 at Baseline
Description: FIB-4 was a noninvasive assessment of liver disease assessed by a combination of age, ALT and platelet results. FIB-4 was the ratio of age in years and aminotransferase to platelet count. It was a non-invasive hepatic fibrosis index score combining standard biochemical values, platelets, ALT, AST and age that was calculated using formula: FIB-4 = (Age [years] x AST [U/L]) / (platelets [10^9/L] x (square root of ALT [U/L])). A FIB-4 index of <1.45 indicated no or moderate fibrosis and an index of > 3.25 indicated extensive fibrosis/cirrhosis. Higher ratio indicated worse condition. Baseline was defined as the last value collected prior to the first administration of the IP.
Time Frame: Baseline (Day 1)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | DB: Placebo | DB: OCA 10 Milligrams (mg) | DB: OCA 10 mg Titrated to OCA 25 mg
Number analyzed (Participants) | 311 | 295 | 308
Ratio | 2.279 (1.1091) | 2.475 (1.9307) | 2.405 (1.1630)

9. Secondary Outcome: DB Phase: ELF at Baseline
Description: ELF was non-invasive panel of circulating fibrosis markers calculated from serum biomarkers. The markers of fibrosis comprised HA, TIMP1 and PIIINP. Each of these markers was measured by an immunoassay and an ELF score was generated, from which a level of fibrosis severity could be determined. The ELF test was a composite score: < 7.7: no to mild fibrosis; ≥ 7.7 - < 9.8: Moderate fibrosis; ≥ 9.8 - < 11.3: Severe fibrosis; ≥ 11.3: Cirrhosis.; higher ELF scores were associated with worsening liver fibrosis. Baseline was defined as the last value collected prior to the first administration of the IP.
Time Frame: Baseline (Day 1)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DB: Placebo | DB: OCA 10 Milligrams (mg) | DB: OCA 10 mg Titrated to OCA 25 mg
Number analyzed (Participants) | 307 | 294 | 307
Scores on a scale | 10.50 (0.921) | 10.60 (0.920) | 10.61 (0.867)

10. Primary Outcome: OLE Phase: Number of Participants With Adjudicated Liver Related Clinical Outcomes: Ascites, Hepatocellular Carcinoma (HCC) and Non-liver Related Death
Description: Adjudication was performed under the review of Hepatic Safety Adjudication Committee (HSAC) of all available data for each identified participant to determine liver injury status. Number of participants with adjudicated liver related clinical outcomes for the following is presented: Ascites (secondary to cirrhosis and requiring medical intervention), Hepatocellular carcinoma (HCC) and non-liver related death.
Time Frame: Up to 12 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Number analyzed (Participants) | 231 | 221 | 207
Participants
  Ascites (secondary to cirrhosis and requiring medical intervention) | 1 | 0 | 2
  HCC | 3 | 1 | 1
  Non-liver related death | 1 | 0 | 1

11. Primary Outcome: OLE Phase: Number of Participants With Adjudicated Liver Related Clinical Outcomes: Worsening of Child-Pugh Score
Description: The Child-Pugh classification was a scoring system used for the classification of the severity of cirrhosis. It included three continuous variables (bilirubin, albumin, and international normalized ratio) and two discrete variables (ascites and encephalopathy). Each variable was scored 1-3 with 3 indicating most severe derangement. The determination of Child-Pugh score ranged from 5 to 15. The higher the score, the sicker the participant. Adjudication was performed under the review of HSAC of all available data for each identified participant to determine liver injury status. Number of participants with adjudicated liver related clinical outcomes for worsening of Child-Pugh score is presented.
Time Frame: Up to 12 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Number analyzed (Participants) | 231 | 221 | 207
Participants | 0 | 1 | 2

12. Primary Outcome: OLE Phase: Number of Participants With Adjudicated Liver Related Clinical Outcomes: Model for End-Stage Liver Disease (MELD) Score ≥15
Description: MELD was a scoring system for assessing the severity of chronic liver disease and to assess prognosis and suitability for liver transplantation. It uses the participant's values for total bilirubin, serum creatinine, and the international normalized ratio for prothrombin time to predict survival. MELD score ranges from 6 (less ill) to 40 (gravely ill) with scores and mortality probability being: Score 40=71.3% mortality; Scores 30-39=52.6% mortality; Scores 20-29=19.6% mortality; Scores10-19=6.0% mortality; Score 9 or less=1.9% mortality. Higher scores indicated greater disease severity. Adjudication was performed under the review of HSAC of all available data for each identified participant to determine liver injury status. Number of participants with adjudicated liver related clinical outcomes for MELD score ≥15 is presented.
Time Frame: Up to 12 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
Number analyzed (Participants) | 231 | 221 | 207
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 18 months for DB phase and Up to 1 year for OLE phase
Description: Safety Population: included all randomized participants who received at least 1 dose of investigational product (OCA or placebo). 3 participants from ITT Population did not receive study treatment, hence were not included in Safety Population.
Arm/Group | DB: Placebo | DB: OCA 10 Milligrams (mg) | DB: OCA 10 mg Titrated to OCA 25 mg | OLE: OCA 10 mg (DB Placebo) | OLE: OCA 10 mg (DB OCA 10 mg) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg)
All-Cause Mortality (participants affected / at risk) | 4/312 | 3/295 | 3/309 | 1/231 | 0/221 | 1/207
Serious Adverse Events (participants affected / at risk) | 43/312 | 49/295 | 46/309 | 26/231 | 50/221 | 48/207
Other Adverse Events (participants affected / at risk) | 290/312 | 276/295 | 291/309 | 199/231 | 213/221 | 197/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=312) | DB: OCA 10 Milligrams (mg) (N=295) | DB: OCA 10 mg Titrated to OCA 25 mg (N=309) | OLE: OCA 10 mg (DB Placebo) (N=231) | OLE: OCA 10 mg (DB OCA 10 mg) (N=221) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg) (N=207)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0 | 2 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 6 | 8
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cryptitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 1 | 2 | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Event leading to Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Granuloma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemobilia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 2 | 3 | 3 | 2 | 7
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 2
COVID-19 (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 3
Campylobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cryptococcal fungaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Endocarditis enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 0 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0
Posterior tibial tendon dysfunction (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 2 | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 2 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Extramammary Paget's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 1 | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Meningoradiculitis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary dissease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=312) | DB: OCA 10 Milligrams (mg) (N=295) | DB: OCA 10 mg Titrated to OCA 25 mg (N=309) | OLE: OCA 10 mg (DB Placebo) (N=231) | OLE: OCA 10 mg (DB OCA 10 mg) (N=221) | OLE: Titrated to OCA 25 mg (DB OCA 10 mg Titrated to OCA 25 mg) (N=207)
Nausea (Gastrointestinal disorders) | 43 | 32 | 48 | 19 | 28 | 39
Constipation (Gastrointestinal disorders) | 20 | 28 | 33 | 12 | 26 | 28
Abdominal pain (Gastrointestinal disorders) | 20 | 31 | 24 | 10 | 25 | 22
Abdominal pain upper (Gastrointestinal disorders) | 29 | 30 | 23 | 12 | 31 | 18
Diarrhoea (Gastrointestinal disorders) | 38 | 28 | 22 | 12 | 24 | 20
Abdominal distension (Gastrointestinal disorders) | 21 | 24 | 23 | 4 | 22 | 21
Vomiting (Gastrointestinal disorders) | 18 | 20 | 25 | 11 | 14 | 21
Varices oesophageal (Gastrointestinal disorders) | 21 | 19 | 21 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 5 | 12
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 9 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 7 | 10
Fatigue (General disorders) | 35 | 27 | 36 | 15 | 27 | 27
Oedema peripheral (General disorders) | 0 | 0 | 0 | 6 | 13 | 16
Urinary tract infection (Infections and infestations) | 29 | 44 | 27 | 13 | 38 | 31
Upper respiratory tract infection (Infections and infestations) | 22 | 19 | 18 | 9 | 23 | 23
Sinusitis (Infections and infestations) | 18 | 20 | 19 | 7 | 22 | 21
Nasopharyngitis (Infections and infestations) | 21 | 13 | 15 | 6 | 20 | 12
Bronchitis (Infections and infestations) | 22 | 14 | 9 | 6 | 13 | 10
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 7 | 21 | 31
Low density lipoprotein increased (Investigations) | 5 | 34 | 33 | 11 | 31 | 17
Blood bilirubin increased (Investigations) | 11 | 14 | 17 | 7 | 14 | 12
Blood creatinine increased (Investigations) | 10 | 14 | 13 | 8 | 19 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 9 | 18 | 21 | 8 | 17 | 21
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 17 | 22 | 7 | 15 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 6 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 22 | 28 | 15 | 24 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 19 | 18 | 6 | 21 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 12 | 16 | 1 | 18 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 17 | 7 | 4 | 17 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 6 | 10
Headache (Nervous system disorders) | 26 | 16 | 20 | 15 | 19 | 21
Dizziness (Nervous system disorders) | 10 | 14 | 14 | 6 | 15 | 12
Insomnia (Psychiatric disorders) | 14 | 16 | 10 | 3 | 16 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 19 | 6 | 14 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 12 | 1 | 8 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 98 | 120 | 177 | 72 | 97 | 120
Rash (Skin and subcutaneous tissue disorders) | 14 | 10 | 29 | 14 | 15 | 23
Hypertension (Vascular disorders) | 0 | 0 | 0 | 8 | 11 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators must wait 18 months after the study ends to publish their results and a multi-center publication must come first. The sponsor has a 45-day review period with the option to extend to an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT03439254/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03439254/SAP_001.pdf